CLINICAL TRIAL: NCT04294706
Title: Effects of Hemp Oil on Markers of Optimal Wellness, Stress Resilience and Recovery in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CVSI-001-2018
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Sleep; Stress; Mood

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemp arm (Experimental): Randomly assignment to Hemp arm (60 mg/day of hemp oil extract x 6 weeks)
  Interventions: Dietary Supplement: Hemp arm
- Placebo arm (Placebo Comparator): Randomly assigned to Placebo arm (60 mg/day of cellulose x 6 weeks)
  Interventions: Dietary Supplement: Hemp arm

INTERVENTIONS:
Dietary Supplement: Hemp arm — Hemp oil

SUMMARY:
The purpose of this placebo-controlled, double-blind study is to determine the effects of a commercially available (i.e. dietary supplement) Hemp Oil Extract product on various markers of physical and mental stress resilience, and perceived recovery from normal daily physical & mental stress. Secondary purposes are to collect information on perceived appetite, mood, feelings of wellbeing, sleep quality, body composition and safety information via standard clinical chemistry panels of sera and plasma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects provide written and dated informed consent to participate in an IRB approved study.
* Subjects are in good health as determined by medical history and routine blood chemistries.
* Subjects are male or female between the ages of 18 and 55 (inclusive).
* Female subjects must agree to use barrier contraceptive methods during sexual intercourse for the duration of the study. All females will undergo pregnancy testing (urine HCG screen) before being screened and at each visit unless they present evidence of surgical sterilization by tubal ligation, bilateral oophorectomy or hysterectomy.
* Subjects have a Body Mass Index of 25-35.
* Subjects are willing and able to comply with the daily activity and supplement protocol.
* Subject is willing and able to comply with the visit schedule.
* Subjects are normotensive (resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg), have a normal resting heart rate (<90 per minute).

Exclusion Criteria:

* Subjects that currently exercise more than three times per week.
* Subject has used weight loss medications within the past three months of Screening visit.
* Subject is on thyroid medication at a dose that is not considered stable. Stable is defined as using the same dose consistently for at least 90 days.
* Subjects with any metabolic disorder including known electrolyte abnormalities, diabetes (or fasting glucose ≥126 mg/dL at the screening visit), unstable or unmanaged thyroid disease, or hypogonadism.
* Subjects with a history of hepato-renal, musculoskeletal, autoimmune, neurologic disease, or any other medical condition deemed exclusionary by the medical staff.
* Subjects taking anti-anxiety, anti-depressant, psychotropic hyperlipidemic, hypoglycemic, anti-coagulant or androgenic medications; nitrates/nitrate derivatives, and PDE-5 inhibitors; and other vasodilatory agents such as calcium channel blockers and beta blockers.
* Subject has an active gastrointestinal disorder such as peptic ulcer disease or malabsorption syndrome (mild lactose intolerance or gastroesophageal reflux diseases are acceptable).
* Subjects who have taken anabolic steroids, growth hormone, IGF-1 or other anabolic drugs within the past year.
* Subjects who are pregnant, trying to become pregnant, or who are nursing.
* Female participants who are < 120 days postpartum before enrolling.
* Subjects who have taken any nutritional supplements that may affect sleep, mood or healthy stress response (including but not limited to Ashwagandha, Valerian root, Melatonin, L-theanine, 5-HTP), or that may affect anabolic/catabolic hormone levels (e.g., androstenedione, DHEA, etc.) within four weeks prior to the start of the study.
* Subjects who have gained or lost more than 5 lbs within 30 days prior to the start of the study.
* Subjects with history of heart disease, peripheral vascular disorders or vaso-occlusive or vasospastic syndromes, psychiatric disorders, or history of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin.
* Subject has a recent history of (within 3 months of Screening Visit) or strong potential for alcohol or substance abuse. Alcohol abuse defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Subject has been hospitalized within the past one-year for any mental or emotional illness.
* Subject has an active infection or sign/symptoms of an infection.
* Subject has dietary tendencies that may be representative of disordered eating (in the opinion of the Investigator).
* Subjects who had any known allergy to any of the ingredients in any of the test products.
* Subjects who are participating in other research studies.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.
* Subjects who smoked or used any tobacco or nicotine containing products within the past year.
* Subjects with syndromes or prescribed medications that may influence body composition, or CVD (e.g. prednisone, Ritalin, Adderall, GH); also protease inhibitors/antivirals (nucleic acid analogs).
* Subjects with orthopedic limitations or injuries that would preclude them from the physical activity intervention in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Sleep quality | baseline
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Sleep quality | week 3
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Sleep quality | week 6
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Stress | Baseline
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Stress | Week 3
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Stress | Week 6
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Well-being | Baseline
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Well-being | Week 3
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Well-being | Week 6
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Readiness to perform exercise | Baseline
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Readiness to perform exercise | Week 3
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Readiness to perform exercise | Week 6
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Appetite | Baseline
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Appetite | Week 3
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Appetite | Week 6
  A visual analog scale constructed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings.
Body composition | Baseline
  DXA measurement
Body composition | Week 3
  DXA measurement
Body composition | Week 6
  DXA measurement

SECONDARY OUTCOMES:
Blood pressure | Baseline
  Measured in mm Hg
Blood pressure | Week 3
  Measured in mm Hg
Blood pressure | Week 6
  Measured in mm Hg
Plasma liver enzyme | Baseline
  Alanine aminotransferase
Plasma liver enzyme | Week 3
  Alanine aminotransferase
Plasma liver enzyme | Week 6
  Alanine aminotransferase
Plasma liver enzyme | Baseline
  Aspartate aminotransferase
Plasma liver enzyme | Week 3
  Aspartate aminotransferase
Plasma liver enzyme | Week 6
  Aspartate aminotransferase
Plasma Lipid panel | Baseline
  Total cholesterol, LDL, HDL and triglycerides
Plasma Lipid panel | Week 3
  Total cholesterol, LDL, HDL and triglycerides
Plasma Lipid panel | Week 6
  Total cholesterol, LDL, HDL and triglycerides

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lopez HL, Cesareo KR, Raub B, Kedia AW, Sandrock JE, Kerksick CM, Ziegenfuss TN. Effects of Hemp Extract on Markers of Wellness, Stress Resilience, Recovery and Clinical Biomarkers of Safety in Overweight, But Otherwise Healthy Subjects. J Diet Suppl. 2020;17(5):561-586. doi: 10.1080/19390211.2020.1765941. Epub 2020 May 27. PMID 32456572